CLINICAL TRIAL: NCT06521125
Title: Clinical Genetics and Screening for Idiopathic Pulmonary Fibrosis
Acronym: GENESI
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RICHELDI LUCA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6869
Record Dates: First submitted 2024-07-16; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Familial Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Respiratory Function Tests; Sequence Analysis, DNA

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with FPF and sporadic IPF
  Interventions: Diagnostic Test: High resolution Computed Tomography (HRCT) scans of the Chest; Diagnostic Test: Pulmonary Function Testing (PFTs); Diagnostic Test: Digital lung sounds auscultation; Diagnostic Test: Laboratory Assessments; Genetic: DNA sequencing
- First-degree relatives of patients with FPF and sporadic IPF
  Interventions: Diagnostic Test: High resolution Computed Tomography (HRCT) scans of the Chest; Diagnostic Test: Pulmonary Function Testing (PFTs); Diagnostic Test: Digital lung sounds auscultation; Diagnostic Test: Laboratory Assessments; Genetic: DNA sequencing

INTERVENTIONS:
Diagnostic Test: High resolution Computed Tomography (HRCT) scans of the Chest — A chest high-resolution computed tomography (HRCT) scan will be performed
Diagnostic Test: Pulmonary Function Testing (PFTs) — Spirometry and diffusing capacity of the lung for carbon monoxide (DLCO) measurements will be performed
Diagnostic Test: Digital lung sounds auscultation — Lung sounds will be recorded using a manual approach with a digital stethoscope
Diagnostic Test: Laboratory Assessments — Clinical laboratory tests will be collected from each participant
Genetic: DNA sequencing — A sample of genomic DNA from peripheral blood lymphocytes will be collected for DNA sequencing

SUMMARY:
Background:

Idiopathic pulmonary fibrosis (IPF) is the most common and severe form of interstitial lung disease. Between 2% and 20% of patients with IPF have a family history of the disease, which is considered the strongest risk factor. Therefore, genetic testing has been increasingly considered as a potential tool to identify patients at risk of developing IPF.

According to some studies, genetic testing (particularly of MUC5B and TERT mutations) could be useful to rapidly identify unidentified and/or asymptomatic individuals (in families as well as in the general population) who have interstitial lung anomalies (ILA) that may indicate a initial stage of pulmonary fibrosis. Finding efficient screening methods and associated targeted treatments for IPF may be essential to improving the prognosis and quality of life of those suffering from this disease.

Objectives of the study:

The study involves two populations of study subjects:

* patients with FPF and sporadic IPF
* first-degree relatives of patients with FPF and sporadic IPF (biological relatives, not spouses)

The primary objective is to determine the prevalence rates of interstitial lung abnormalities in at-risk relatives of patient with IPF and FPF.

Study design:

Multicenter, cross-sectional study without drug and without device conducted in two major Italian tertiary referral hospitals.

The entire project is expected to last 24 months.

ELIGIBILITY:
Criteria for PATIENTS:

Inclusion Criteria:

1. patients aged ≥18 years when signing the informed consent
2. diagnosis of IPF based on 2022 ATS/ERS/JRS/ALAT Guidelines as confirmed by the investigator based on chest HRCT scan and if available surgical lung biopsy
3. diagnosis of FPF defined as the presence of fibrotic ILD in at least two members of the same biological family
4. at least one 1st degree relative >40 years of age.

Exclusion Criteria:

1. patients with Interstitial Lung Diseases other than Idiopathic Pulmonary Fibrosis, including but not limited to patients with granulomatous lung disease, autoimmune/collagen vascular disease associated interstitial lung disease, and drug induced interstitial lung disease
2. unwilling or unable to sign informed consent

Criteria for FIRST DEGREE BIOLOGICAL RELATIVES:

Inclusion Criteria:

a. subjects aged ≥40 years

Exclusion Criteria:

1. previous diagnosis of IPF
2. a history of severe or poorly controlled anxiety, severe or poorly controlled depression according to the opinion of the investigators, suicidal ideation, or other psychiatric illness requiring hospitalization
3. unwilling or unable to sign informed consent 400 first-degree relatives of participating patients will be recruited

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study involves two populations of study subjects:
  * patients with FPF and sporadic IPF
  * first-degree relatives of patients with FPF and sporadic IPF (biological relatives, not spouses).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of ILA | At subject enrollment
  The prevalence of ILA in first-degree relatives of patients with IPF, expressed as proportion of subjects with ILAs in the overall relatives population

SECONDARY OUTCOMES:
Association between ILA and genetic variants | At subject enrollment
  To assess the risk of ILA in first-degree relatives of patients with FPF and sporadic IPF associated with clinically relevant mutations.
  Univariate and multivariate logistic regression analysis will be utilized to assess the association between genetic variants and ILA